CLINICAL TRIAL: NCT06615089
Title: Effect Of Balance Training With Foot Orthosis On Falling In Elderly
Acronym: FO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Youmn Nabil Saad Zaghloul Hafez, principal investigator youmn nabil saad zaghloul, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/004445
Record Dates: First submitted 2024-09-24; First posted 2024-09-26 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Elderly
Keywords: balance trainig; foot orthosis; elderly

STUDY DESIGN:
Intervention Model Description: balance training and foot orthosis
Who Masked: Outcomes Assessor
Masking Description: opaque sealed envelope
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- balance training (Experimental): thirty elderly patients will receive balance training and orthotic prescription for four months
  Interventions: Other: balance training; Other: orthotic prescription
- orthotic prescription (Active Comparator): thirty elderly patients will receive orthotic prescription for four months
  Interventions: Other: orthotic prescription

INTERVENTIONS:
Other: balance training — the elderly patients will receive balance training in the form of proprioceptive and vestibular training components. proprioceptive training include Standing static balance, lateral weight transfer, Lateral weight transfer near to chair, tandem closed eyes, walking on toes, Postural control using ball. Vestibular training in the form of Balance with head movement, seated lateral step in addition to Insoles inside the subjects' own regular shoes
  Arms: balance training
Other: orthotic prescription — the elderly patients will receive Insoles inside the subjects' own regular shoes

SUMMARY:
this study will be conducted to investigate effect of balance training with foot orthosis on falling in elderly.

DETAILED DESCRIPTION:
The concept of physiology of ageing implies that a series of complex events occur which ultimately lead to a progressive reduction in function of all organ systems. This process, also called "homeostenosis," is influenced by gene variations and differences in exposure to environmental factors .Reduction in muscle strength and coordination of the lower extremities accompanied by decreased gait assurance and balance control are the result of a physical deterioration in an older body. Together with decreased cognitive functions, these impairments lead to a higher risk of falling among the elderly. The foot is the first point of contact between the body and the external environment, and it plays an important role in postural sway. Its plantar mechanical receptors provide spatial and temporal information about contact pressures and shear forces resulting from body movement being a valuable feedback mechanism to the postural control system. Interventions to optimize sensory information from plantar sole such as vibration stimuli, customized foot orthoses, textured insoles, and sandals with textured insoles and magnetic insoles have been tested before, some of them showing balance improvement .Sixty elderly patients will be allocated randomly to two groups; group 1 will receive balance training program beside orthotic prescription and group 2 will receive orthotic prescription alone.

ELIGIBILITY:
Inclusion Criteria:

* Age 65-75years
* Both gender
* Body mass index 25-29.9 kg/m2
* All participants will use foot orthosis
* Clinically and medically stable patients
* having a Berg Balance Scale (BBS) score between 35 and 45
* Scored 19-21 will be regarded as being at moderate risk of falling,
* Scored 19-23 in the Tinetti tool score
* Scored more than 13.5 sec in timed up-and-go test

Exclusion Criteria:

* Bedridden subjects.
* Previous vestibular diseases, central nervous system pathologies (such as stroke, dementia, Parkinson, etc.).
* Previous diagnosis of peripheral neuropathy.
* current use of medications affect the result of the study
* Use of insoles in the last month
* Previous history of foot surgery, and amputation of the lower limbs.
* severe foot deformity (not able to wear regular shoes), difficulty in adapting insoles inside his/her own shoes,
* Patient with life threatening disorders as renal failure, myocardial infarction.
* Patients who suffering from myasthenia gravis, hyperthyroidism, haemorrhage, acute viral disease, acute tuberculosis, mental disorders or those with pacemakers.
* Un controlled diabetes, hypertension and smokers

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
balance | up to four months
  The Berg Balance Scale (BBS) will be used to assess balance. it measure the ability of a subject to maintain balance while performing 14 movements required in everyday activities . Scoring is based on an ordinal 5-point scale of 0 to 4. A score of 0 is given if the subject is unable to complete the task and a 4 is given if the subject is able to complete the task unassisted. The maximum possible score is 56

SECONDARY OUTCOMES:
gait assessment | up to four months
  The Dynamic gait index was primarily developed to assess a subject's ability to modify gait in response to changing task demands.The eight abilities assessed are: steady-state walking, walking while changing gait speed, walking while moving the head vertically and horizontally, walking while stepping over and around an obstacle, pivoting during walking, and stair climbing. The items of the DGI are graded on a four-point scale from 'normal performance' (3) to 'severely impaired' (0), yielding a maximum score of 24 points
balance deficit | up to four months
  The Timed "up and go" test is performed in the following way. The patient will sit on a standard arm chair (seat height 46cm as in the original setting, arm height 67cm) with his or her back against the chair, arms resting on the chair's arms and walking aid at hand. Patients will wear their regular footwear and will use their customary walking aids. After the patient will state that he or she is ready, the test will start. On the word "go" the patient will stand, will walk to a line on the floor 3m away (on a standard short-piled carpet with a length of 4m and width of lm), turns, will walk back to the chair, and will sit down again.
gait and balance assessment | up to four months
  The Tinetti Assessment Tool is a simple test that measures a participant's gait and balance. The participant performs a total of 16 tasks (during 9 tests the researcher assesses the balance of the participant and during 7 subsequent tests the researcher assesses the gait of the participant). Scoring of the Tinetti Assessment Tool is done on a two or 3-point ordinal scale (depending on the task) with a range of 0 to 1 or 0 to 2. A score of 0 represents the most impairment, while a score of 1 or 2 represents independence